CLINICAL TRIAL: NCT03405688
Title: Transfusion in Sickle Cell Disease: Screening of Sickle Cell Disease Trait in Blood Donors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanane EL KENZ (Other)
Responsible Party: Sponsor-Investigator, Hanane EL KENZ, Head of Blood Bank, Brugmann University Hospital
Organization: Brugmann University Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUB-PRO-TRANSFU-DREPANO 2
Record Dates: First submitted 2018-01-15; First posted 2018-01-23 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Sickle Cell Disease; Sickle Cell Trait
Keywords: Sickle cell; Heterozygous; Blood donor
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Acute transfusion (Experimental): Blood donor heterozygous for the sickle cell disease allele (HbAS genotype)
  Interventions: Procedure: Blood sampling
- Control - Acute transfusion (Other): Blood donor not bearer of the sickle cell disease allele (HbAA genotype)
  Interventions: Procedure: Blood sampling
- Chronic transfusion (Experimental): Blood donor heterozygous for the sickle cell disease allele (HbAS genotype)
  Interventions: Procedure: Blood sampling
- Control - Chronic transfusion (Other): Blood donor not bearer of the sickle cell disease allele (HbAA genotype)
  Interventions: Procedure: Blood sampling
- Transfusion prior to surgery (Experimental): Blood donor heterozygous for the sickle cell disease allele (HbAS genotype)
  Interventions: Procedure: Blood sampling
- Control - Transfusion prior to surgery (Other): Blood donor not bearer of the sickle cell disease allele (HbAA genotype)
  Interventions: Procedure: Blood sampling

INTERVENTIONS:
Procedure: Blood sampling — Extra blood samples taken for laboratory analysis

SUMMARY:
Bearers of the sickle cell allele (S) are currently eligible for blood donations in Belgium. As blood donors are not tested for this allele, their heterozygous status is unknown. However, guidelines recommend to transfuse sickle cell patients with blood that is negative for the 'S' hemoglobin. To the investigator's knowledge, no study has been conducted to evaluate the impact of transfusion with blood originating from heterozygous donors on the transfusion performance and the improvement of clinical status of the sickle cell disease patients.

ELIGIBILITY:
Inclusion Criteria:

All patients with sickle cell disease within the CHU Brugmann and the Queen Fabiola Children's Hospital (HUDERF)

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2018-02-13 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin level -patient | 1 hour before blood transfusion
  Hemoglobin level (g/dL)
Hemoglobin level -patient | 1 hour after blood transfusion
  Hemoglobin level (g/dL)
% of 'S' type hemoglobin -patient | 1 hour before blood transfusion
  % of 'S' type hemoglobin (assessed by means of hemoglobin electrophorese)
% of 'S' type hemoglobin -patient | 1 hour after blood transfusion
  % of 'S' type hemoglobin (assessed by means of hemoglobin electrophorese)
Hemoglobin level - transfused blood | 1 hour before blood transfusion
  Hemoglobin level (g/dL)
% of 'S' type hemoglobin -transfused blood | 1 hour before blood transfusion
  % of 'S' type hemoglobin (assessed by means of hemoglobin electrophorese)
Transfusion yield | 1 hour after blood transfusion
  Computed by means of a formula taking the level of hemoglobin, the % of 'S' type hemoglobin and the body surface into account.
Medical complications | 1 month
  List of medical complications having occured after a surgery. Applicable only to the 'transfusion prior to surgery' groups.
Length of stay | 1 month
  Length of stay within the hospital. Applicable only to the 'acute transfusion' groups
Length of stay post transfusion | 1 month
  Length of stay within the hospital after a blood transfusion. Applicable only to the 'acute transfusion' groups
Number of blood transfusions | 1 month
  Number of blood transfusions. Applicable only to the 'acute transfusion' groups
Hospital re-admission | 1 month
  Hospital re-admission. Applicable only to the 'acute transfusion' groups
Mortality rate | 1 month.
  Mortality rate. Applicable only to the 'acute transfusion' groups

CONTACTS AND LOCATIONS:
Overall Officials: Marie Deleers, Ph Biol, Principal Investigator — CHU Brugmann
Locations (2):
- Belgium (2):
  - CHU Brugmann, Brussels
  - HUDERF, Brussels

IPD SHARING:
Plan to Share IPD: No